CLINICAL TRIAL: NCT03680417
Title: Reactogenicity and Protectivity Following Measles- Rubella (MR) Routine Immunization in Indonesian Infants and Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PMS-MR-0417
Record Dates: First submitted 2018-09-18; First posted 2018-09-21 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Safety Issues; Immunogenicity
Keywords: Measles-Rubella; Vaccine; Safety; Immunogenicity; Reactogenicity; Protectivity
MeSH Terms: interventions — Vaccines

STUDY DESIGN:
Intervention Model Description: Safety Group: open labeled, prospective intervention study, only assess the safety outcome Sub Group: open labeled, prospective intervention study, evaluate safety and protectivity outcome
Who Masked: Outcomes Assessor
Masking Description: laboratory analyst are masked for the evaluation of antibody against measles and rubella. The immunogenicity is measured before and after vaccination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safety Study (Measles-Rubella vaccine) (Active Comparator): open labeled, prospective intervention study, only assess the safety outcome. The Measles-Rubella vaccine is administered in infants age 9-12 months or 18 - 47 months. This study group only assessed for safety profile of the Measles-Rubella vaccine.
  Interventions: Biological: Measles-Rubella (MR) Vaccine
- Sub Study (Measles-Rubella vaccine) (Active Comparator): open labeled, prospective intervention study, assess the safety and immunogenicity outcome. The Measles-Rubella vaccine is administered in infants age 9-12 months or 18 - 47 months. For Sub study, pre- and post immunization sera will be obtained from 200 infants and/or children. Safety assessment also evaluated for 28 days after immunization.
  Interventions: Biological: Measles-Rubella (MR) Vaccine

INTERVENTIONS:
Biological: Measles-Rubella (MR) Vaccine — Measles and Rubella Vaccine, live attenuated (Serum Institute of India) Form : Freeze dried Dose : 1 dose 0.5 ml contains not less than 1000 CCID50 of measles virus and 1000 CCID50 of rubella virus.

SUMMARY:
to assess safety and immunogenicity of measles-rubella (MR) routine immunization in Indonesian Children and Infants

DETAILED DESCRIPTION:
* to asses serious immediate systemic events,
* to assess local and systemic reaction after Measles-Rubella (MR) vaccine in infants and children,
* to evaluate protectivity and antibody response to measles and rubella after 1 dose of MR vaccine

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants (9-12 months) or children (18-47 months)
* Will receive MR routine immunization.
* Parents have been informed properly regarding the study and signed the informed consent form.
* Parents will commit themselves to comply with the instructions of the investigator and the schedule of the trial.

Exclusion Criteria:

* MR vaccine given simultaneously with other vaccination, except Pentabio (DTP/HB/Hib)

Ages: 9 Months to 47 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 590 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2018-02-26 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Number of Immediate systemic events | 30 minutes
  Number of subjects with at least one serious immediate systemic events within 30 minutes after vaccination
Percentage of immediate systemic events | 30 minutes
  Percentage of subjects with at least one serious immediate systemic events within 30 minutes after vaccination

SECONDARY OUTCOMES:
Local reaction | 72 hours
  Number of subjects with at least one local reaction occurring within 72 h after vaccination.
Systemic reaction | 72 hours
  Number of subjects with at least one systemic event occurring within 72 h after vaccination.
Delayed Local reaction | 11 days
  Number of subjects with at least one local reaction occurring between day 4-14 after vaccination.
Delayed systemic event | 11 days
  Number of subjects with at least one systemic event occurring between day 4-14 after vaccination.
Late Local reaction | 14 days
  -Number of subjects with at least one systemic event occurring between day 15 to 28 following vaccination.
Late Safety (Systemic event) | 14 days
  Number of subjects with at least one systemic event occurring between day 15 to 28 following vaccination.
Safety (serious adverse event) | 28 days
  - Number of serious adverse event occuring from inclusion until 28 days after immunization
Immunogenicity for Measles (subject with anti measles titer ≥ 8 (1/dil)) | 28 days
  - Percentage of subjects with anti measles titer ≥ 8 (1/dil), 28 days after one dose of MR vaccine in Infants & Children.
Immunogenicity for Measles (Geometric Mean Titer) | 28 days
  - Geometric Mean Titer of measles antibody
Immunogenicity for Measles (increasing measles antibody titer ≥ 4 times) | 28 days
  - Percentage of infants with increasing measles antibody titer ≥ 4 times
Immunogenicity for Measles (seroconversion from seronegative to seropositive) | 28 days
  - Percentage of infants with transition of seronegative to seropositive.
Immunogenicity for Rubella (Subjects with anti rubella titer ≥11 IU/ml) | 28 days
  - Percentage of subjects with anti rubella titer ≥11 IU/ml, 28 days after one dose of MR vaccine in Infants & Children.
Immunogenicity for Rubella (Geometric Mean Titer) | 28 days
  - Geometric Mean Titer of Rubella antibody.
Immunogenicity for Rubella (increasing rubella antibody titer ≥ 4 times) | 28 days
  - Percentage of infants with increasing rubella antibody titer ≥ 4 times
Immunogenicity for Rubella (seroconversion from seronegative to seropositive) | 28 days
  - Percentage of infants with transition of seronegative to seropositive.

CONTACTS AND LOCATIONS:
Overall Officials: Dominicus Husada, Dr, Principal Investigator — Child Health Dept. Dr. Soetomo Hospital/School of Medicine, Airlangga Univ.
Locations (1):
- Child Health Dept. Dr. Soetomo Hospital, School of Medicine Airlangga Univ., Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No